CLINICAL TRIAL: NCT01404663
Title: Evaluation the Side Effects of Bone Marrow Derived CD133 Cells Transplantation in Cerebral Palsy Patients
Brief Title: Side Effects of Bone Marrow Derived CD133 Transplantation in Cerebral Palsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-nerve-002
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2010-08

CONDITIONS: Cerebral Palsy
Keywords: bone marrow CD133 transplantation side effects; side effects
MeSH Terms: conditions — Cerebral Palsy | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell recipients (Experimental): The 4-12 years old patients with cerebral palsy who undergone bone marrow derived CD133 transplantation
  Interventions: Biological: CD133 stem cell injection

INTERVENTIONS:
Biological: CD133 stem cell injection — Bone marrow derived CD133 stem cell witch are transplanted by intrathecal injection
  Other Names: stem cell transplantation

SUMMARY:
Cerebral palsy (CP) is condition, sometimes thought of as a group of disorders that can involve brain and nervous system functions such as movement, learning, hearing, seeing, and thinking.Cerebral palsy is caused by injuries or abnormalities of the brain. Most of these problems occur as the baby grows in the womb, but they can happen at any time during the first 2 years of life, while the baby's brain is still developing.Bone marrow derived stem cells are known as a effective therapy.

In this study the investigators evaluate the side effect of bone marrow stem cell transplantation in patients with cerebral palsy.

DETAILED DESCRIPTION:
Our study evaluate the side effects of bone marrow derived CD133 cells transplantation in 4-12years old patients with cerebral palsy.first all the patients undergone a comprehensive evaluation(physical exam, serology tests,EEG,MRI,GMFM66).

After bone marrow aspiration,autologous stem cells prepare for each patient. In operation room ,the cells are transplanted by intrathecal injection. all the patients would be under observed to notice acute side effects and 3,6,9 and 12 months after injection they will be followed and evaluate by comprehensive tests.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of spastic quadriplegic CP
2. Children must be between the ages of 4 and 12 years
3. Children must be cleared by an orthopedic surgeon for risk of hip subluxation or dislocation and cannot have significant scoliosis (curvature > 40 degrees)
4. Children must be seizure-free or seizure controlled

Exclusion Criteria:

1. Children who have a diagnosis of "mixed" types of CP (i.e. athetosis) or other movement disorders (i.e. ataxia)
2. Children who have had a selective dorsal rhizotomy, are presently are receiving intrathecal Baclofen, or have changed their spasticity medications in the past 6 months.
3. Children who have a metallic or electrical implants

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
allergic reaction | 1 month
  evaluation the side effects of bone marrow derived CD133 transplantation in cerebral palsy patients
local infection | 1 month
  infections in site of injection
encephalitis | 1 month
  encephalitis due to cell transplantation
meningitis | 1 month
  meningitis due to cell trnsplantation
paralysis or sensory loss | 6 months
  paralysis or sensory loss below the level of the injection site

SECONDARY OUTCOMES:
speech | 6 months
  evaluation the effect of bone marrow derived CD133 cells transplantation to improve speech ability in patients with cerebral palsy
motion | 6 months
  evaluation the effect of bone marrow derived CD133 transplantation to improve motion disability in patients with cerebral palsy

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Cell therapy Center; AliReza Zaali, MD, Principal Investigator — Head of Research center of neurosurgery; Leila Arab, MD, Principal Investigator — Department of regenerative medicine,Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Zali A, Arab L, Ashrafi F, Mardpour S, Niknejhadi M, Hedayati-Asl AA, Halimi-Asl A, Ommi D, Hosseini SE, Baharvand H, Aghdami N. Intrathecal injection of CD133-positive enriched bone marrow progenitor cells in children with cerebral palsy: feasibility and safety. Cytotherapy. 2015 Feb;17(2):232-41. doi: 10.1016/j.jcyt.2014.10.011. Epub 2014 Nov 1. PMID 25593079
- See also: Related Info — http://Royaninstitute.org